CLINICAL TRIAL: NCT05769543
Title: Impact of WATSU on Body Awareness
Brief Title: WATSU and Body Awareness
Acronym: IWOBA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johannes Kepler University of Linz (Other)
Collaborators: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: IWOBA_1
Record Dates: First submitted 2023-03-03; First posted 2023-03-15 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2023-03

CONDITIONS: Perception, Self; Body Image; Self-Assessment
Keywords: Body Awareness; WATSU

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- WATSU application (Active Comparator)
  Interventions: Procedure: WATSU application
- Control (Placebo Comparator)
  Interventions: Other: Lecture

INTERVENTIONS:
Procedure: WATSU application — 20-minute application of WATSU
  Arms: WATSU application
Other: Lecture — 20-minute lecture on WATSU technique
  Arms: Control

SUMMARY:
Body awareness (BA) is an essential factor for health and well-being. In 2021, the IOBA (Impact on Body Awareness) study was conducted at the Institute of Physical Medicine & Rehabilitation at Kepler University Hospital. Thereby, the impact of massage and of gymnastics on BA in healthy individuals was surveyed. The protocol provides a solid basis for further research projects on BA. In the present study, the direct effect of a WATSU® (Shiatsu in Water) application on BA as well as on the state of health of healthy persons will be determined and BA will be further investigated.

In a randomized controlled study with 60 healthy adults in two groups (WATSU and control group), the use of the Awareness Body Chart (ABC) questionnaire and further German questionnaires (Short questionnaire on self-perception of the body, self-rating mood scale - revised) concerning body awareness and well-being should analyse the following hypothesis: There is a difference in the change of BA between the WATSU group and the control group. Before interventions demographic data and further questionnaires concerning health conditions of the participants (Simple Physical Activity Questionnaire, Short Form Health Survey, Brief Symptom Inventory, Like/Dislike Body Chart and additional questions) are administered. Correlations between BA and the results of these tests will be investigated too. All these analyses can provide innovative information about BA and be indicative in the use of physiotherapeutic measures.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Signing of informed consent by participants and head of the study
* Understanding of German language in order to be able to follow a lecture and complete questionnaires

Exclusion Criteria:

* Current sick leave
* Pregnancy
* Acute physical or psychological complaints on the day of study participation
* Chronic illnesses / disabilities which contraindicate participation or make it difficult to use the therapy pool
* Current illnesses or injuries

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-03-20 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Awareness Body Chart Questionnaire | Before intervention
  Body charts to fill in with colours according to intensity of body awareness. In sum, 51 body regions to colour with 5 different colour pencils (orange = "I can perceive with much detail", yellow = "I can perceive distinctly", green = "I can perceive", blue = "I can perceive indistinctly", black = "I cannot perceive"). To quantify the information, every region of the body will be coded as an extra item and the data of the colours will be transcribed: orange (= 5), yellow (= 4), green (= 3), blue (= 2), black (= 1). Higher values mean higher intensity of body awareness.
Awareness Body Chart Questionnaire | Immediately after intervention
  Body charts to fill in with colours according to intensity of body awareness. In sum, 51 body regions to colour with 5 different colour pencils (orange = "I can perceive with much detail", yellow = "I can perceive distinctly", green = "I can perceive", blue = "I can perceive indistinctly", black = "I cannot perceive"). To quantify the information, every region of the body will be coded as an extra item and the data of the colours will be transcribed: orange (= 5), yellow (= 4), green (= 3), blue (= 2), black (= 1). Higher values mean higher intensity of body awareness.

SECONDARY OUTCOMES:
Short questionnaire on self-perception of the body | Before intervention
  Verbal questionnaire concerning body awareness. 20 items (5 = "I can perceive with much detail", 4 = "I can perceive distinctly", 3 = "I can perceive", 2 = "I can perceive indistinctly", 1 = "I cannot perceive"). Higher values mean higher intensity of body awareness.
Short questionnaire on self-perception of the body | Immediately after intervention
  Verbal questionnaire concerning body awareness. 20 items (5 = "I can perceive with much detail", 4 = "I can perceive distinctly", 3 = "I can perceive", 2 = "I can perceive indistinctly", 1 = "I cannot perceive"). Higher values mean higher intensity of body awareness.
Self-rating mood scale - revised | Before intervention
  Verbal questionnaire concerning mood status. 24 pairs of oppositional adjectives concerning mood: One of them or <neither nor> should be ticked, depending on how it best corresponds to the current situation. The negative pole = 2. The positive pole = 0. <neither nor> = 1. Higher sum scores indicate worse subjective mood, lower values better mood.
Self-rating mood scale - revised | Immediately after intervention
  Verbal questionnaire concerning mood status. 24 pairs of oppositional adjectives concerning mood: One of them or <neither nor> should be ticked, depending on how it best corresponds to the current situation. The negative pole = 2. The positive pole = 0. <neither nor> = 1. Higher sum scores indicate worse subjective mood, lower values better mood.

OTHER OUTCOMES:
Simple Physical Activity Questionnaire | Before intervention
  Questionnaire to survey physical activity: It should show a snapshot of hours per day of an average day in the past week. The time in bed, the time while doing sedentary work (including dozing), while walking, while exercising and during other physical activities (such as household chores) is interrogated. The test does not measure the intensity of physical activity, but rather sorts it into the groups walking, sport and other categories.
Short Form Health Survey (SF-12) | Before intervention
  Questionnaire on health-related quality of life. It consists of twelve questions relating to the last four weeks and yields statements about eight different dimensions of subjective health: general health perception, physical health, physically-conditioned role function, physical pain, vitality, mental health, emotionally-related role function, social functionality. Different Likert-Scales are used. A physical sum scale and a psychological sum scale can be calculated. The polarity of four items must be reversed so that higher values in all items and total scales reflect a better state of health. Normative data are available.
Brief Symptom Inventory | Before intervention
  Questionnaire on the burden of symptoms. The BSI is also called the Brief Symptom Check List (BSCL), it is a short form of the SCL-90 (Derogatis, 1993). The BSI consists of 53 items (physical as well as psychological symptoms), which are assessed subjectively on a Likert scale in relation to the last seven days from 0 = "not at all" to 5 = "very strong". The items result in nine scales: somatization, obsession-compulsion, interpersonal sensitivity, depression, anxiety, hostility, phobic anxiety, paranoid ideation and psychoticism.
Beck Depression Inventory II (BDI-II) | Before intervention
  The BDI-II represents a self-rating instrument to assess the severity of depression. Four statements are given for each of 21 questions, from which the one that best describes how the person has felt in the past week is to be selected. In scoring, each item is given a score of 0 to 3, depending on the choice (higher number means higher depression scores), and after directly adding the scores of the individual items, a total score of 0 to 63 is obtained.
Body Mass Index | Before intervention
  Relation of body weight to the square of body height
Like/Dislike Body Chart | Before intervention
  As an extension to the ABC, this questionnaire is intended to answer the question of whether there are areas of the body that one particularly likes about oneself or that one dislikes about oneself. If yes, one can draw these with a purple color pencil ("particularly like") and/or with a gray color pencil ("do not like") in an extra Body Chart.
Additional questions | Before intervention
  Questions on demographic data and chronic complaints and current illnesses
Charlson Comorbidity Index | Before intervention
  Questionnaire on comorbidities
Feedback form | Immediately after investigation
  Personal feedback on questionnaires and measures

CONTACTS AND LOCATIONS:
Locations (1):
- Kepler University Hospital, Linz, Austria